CLINICAL TRIAL: NCT02121704
Title: Magnetic Endoscope Imaging in Colonoscopy: Influence on Propofol Dosage
Acronym: MEXICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEXICO
Record Dates: First submitted 2014-04-15; First posted 2014-04-23 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Failed Conscious Sedation During Procedure
Keywords: Sedation; Colonoscopy; Propofol; Scope guide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controll Group (No Intervention): Patients from the control group will be examined using a CF-HQ 190 EVIS Exera III Advanced Diagnostic Video Colonoscope. The Magnetic Endoscope Imaging (Scope Guide) function WILL NOT BE USED during the investigation.
- Intervention (Active Comparator): Patients from the control group will be examined using a CF-HQ 190 EVIS Exera III Advanced Diagnostic Video Colonoscope. The Magnetic Endoscope Imaging (Scope Guide) function WILL BE USED during the investigation.
  Interventions: Device: Magnetic Endoscope Imaging (Scope Guide)

INTERVENTIONS:
Device: Magnetic Endoscope Imaging (Scope Guide)
  Other Names: brand name: Scope guide
  Arms: Intervention

SUMMARY:
Magnetic Endoscope Imaging (MEI) is an optional tool which can be switched on at the beginning of colonoscopy. MEI works by creating an electromagnetic field of very low intensity. By that the position of the endoscope can be displayed virtually on a monitor. The use of MEI has been shown to reduce the formation of loops and to ease the removal of existing loops during the investigation. Furthermore, as loops favour the occurrence of pain when the scope is moved forward, patients who underwent colonoscopy with MEI reported less pain at the end of the procedure.

Sedation is used widely during colonoscopy for it has improved the tolerability of the investigation. Most of the patients demand for sedation. In Germany Propofol is recommended as the first-line sedative when endoscopy it is performed in an outpatient setting. The use of Propofol involves the danger of respiratory complications. One reason for the application of Propofol doses is the occurrence of pain during the investigation. We hypothesized that if MEI is used and if loops can be avoided sufficiently lower Propofol doses would be needed. We therefore planned this prospective controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* medical indication for colonoscopy
* age >18 years
* written consent given by patient
* investigation under sedation with propofol

Exclusion Criteria:

* application of any other sedative than propofol
* age < 18 years
* pregnant women
* patients denying written consent
* ASA class IV, V and VI
* indication for colonoscopy: emergency (e.g. severe rectal bleeding)
* allergy to propofol
* pre-existing hypotension, bradycardia or hypoxemia
* history of sedation accidents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Propofol dose | up to one day (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 1 day)
  At the end of colonoscopy total dose of Propofol applicated will be assessed.

SECONDARY OUTCOMES:
Hypoxemia | up to 1 day (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 1 day)
  Oxygen saturation will be measured for the duration of colonoscopy/hospital stay.
Adenoma detection rate | up to one day

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — II. Medizinische Klinik, Klinikum rechts der Isar der Technischen Universität München, Germany; Stefan von Delius, MD, Study Director — Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, München, Deutschland, Germany

REFERENCES:
- [Derived] Klare P, Hartrampf B, Haller B, Schlag C, Geisler F, Abdelhafez M, Einwachter H, Bajbouj M, Schmid RM, von Delius S. Magnetic endoscope imaging for routine colonoscopy: impact on propofol dosage and patient safety - a randomized trial. Endoscopy. 2016 Oct;48(10):916-22. doi: 10.1055/s-0042-110933. Epub 2016 Jul 21. PMID 27441684